CLINICAL TRIAL: NCT07270042
Title: Evaluation of the Efficacy of Zinc on the Duration and Effictiveness of Botulinum Toxin A Injection in the Context of Hyperactive Masseter Muscle (A Prospective Clinical Study)
Brief Title: Evaluation the Efficacy of Zinc on Botulinum Toxin A Injection
Acronym: BTX-A
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TishreenU maxilofacial surgery
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Hyperactive Masseter Muscle
Keywords: Masseter Muscle; Botulinum Toxin; zinc; electromyographic (EMG)
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution; Zinc

STUDY DESIGN:
Intervention Model Description: patients will be randomized in two groups (test group and control group)
Who Masked: Participant, Care Provider
Masking Description: The investigational pharmacy will prepare identical opaque capsules (zinc or placebo) labeled solely by subject ID and treatment period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zinc arm (Experimental): BTX-A Injection with Zinc
  Interventions: Drug: BOTOX 100U in normal saline with zinc
- Placebo arm (Placebo Comparator): BTX-A Injection with placebo
  Interventions: Drug: BOTOX 100U in normal saline with placebo

INTERVENTIONS:
Drug: BOTOX 100U in normal saline with zinc — Pre-treatment (Period days -4 to -1)
  • Zinc arm: Zinc gluconate 50 mg orally once daily for 4 days prior to injections.
  BTX-A injections (Period day 0)
  * Agent: botulinum toxin A (BTX-A).
  * Target: Bilateral masseter muscles only.
  * Dose and mapping: 25-30 Units per side, delivered at 3 standardized points within the masseter safe zone. Mapping is guided by palpation at maximum voluntary clench (MVC) to identify the hypertrophic belly; injections are placed into the muscle belly, avoiding parotid duct and mandibular notch.
  A washout interval of at least 5-6 months, or until the masseter EMG amplitude returns to ≥80% of baseline, will separate the two treatment phases to eliminate residual BTX-A effects and avoid carryover.
  We reinject (BTX-A) to the same patient , but with a Placebo
  Arms: Zinc arm
Drug: BOTOX 100U in normal saline with placebo — Pre-treatment (Period days -4 to -1)
  • Placebo arm: Identical capsule orally once daily for 4 days prior to injections.
  Adherence is reinforced with written instructions, dosing calendars, and pill counts.
  BTX-A injections (Period day 0)
  * Agent: botulinum toxin A (BTX-A).
  * Target: Bilateral masseter muscles only.
  * Dose and mapping: 25-30 Units per side, delivered at 3 standardized points within the masseter safe zone. Mapping is guided by palpation at maximum voluntary clench (MVC) to identify the hypertrophic belly; injections are placed into the muscle belly, avoiding parotid duct and mandibular notch.
  A washout interval of at least 5-6 months, or until the masseter EMG amplitude returns to ≥80% of baseline, will separate the two treatment phases to eliminate residual BTX-A effects and avoid carryover.
  We reinject (BTX-A) to the same patient , but with zinc
  Arms: Placebo arm

SUMMARY:
This clinical trial seeks to investigate a promising new approach to enhance the effectiveness and duration of Botulinum Toxin A (BTX-A) for the treatment of hyperactive masseter muscles. By investigating the role of oral zinc supplementation, this study could provide a cost-effective, sustainable solution for patients suffering from both aesthetic concerns and functional limitations associated with MMH and bruxism. The findings of this study will expand the clinical applications of BTX-A, offering longer-lasting relief and reducing the need for frequent injections, which could revolutionize the management of MMH in clinical practice.

DETAILED DESCRIPTION:
This study aims to explore the potential for oral zinc supplementation to enhance the efficacy and duration of Botulinum Toxin A (BTX-A) in treating hyperactive masseter muscles (MMH). MMH leads to cosmetic deformities like a "square jaw," and is sometimes associated with bruxism and functional issues. While BTX-A is effective for reducing muscle activity, its effects typically last 2-3 months, requiring frequent re-injections. The study hypothesizes that zinc supplementation, which plays a crucial role in synaptic transmission, may prolong and enhance the effects of BTX-A. The trial will be a randomized, double-blind, two-period design at Lattakia University Hospital, recruiting 20 participants aged 18-60 years, who will be randomly assigned to two treatment sequences.

The intervention protocol includes participants with a clinical diagnosis of MMH (with or without bruxism). They will undergo two separate treatment periods: one with zinc gluconate (50 mg/day for 4 days) followed by BTX-A injection, and the other with an identical placebo followed by the same BTX-A protocol. The two treatment periods will be separated by a 5-6 month washout period to eliminate carryover effects, ensuring that the results of the first treatment phase do not influence the second phase.

The primary outcome will be the percentage change in masseter electromyographic (EMG) amplitude at 12 weeks post-injection, compared with baseline (normalized to maximal voluntary clench [MVC]). This will provide data on the magnitude and duration of BTX-A's effect when combined with zinc supplementation. Secondary outcomes will include pain reduction (measured by the Visual Analog Scale [VAS]), patient satisfaction (assessed by a 5-point Likert scale), and time to recovery (time taken for EMG to return to 80% of baseline levels). Additionally, adverse events such as muscle weakness, asymmetry, and bruising will be monitored.

The results of this research could provide a cost-effective and sustainable solution for MMH patients, improving the duration and efficacy of BTX-A treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants will be adults aged 18-60 years presenting with clinically confirmed masseteric hypertrophy or hyperactivity, as approved by EMG.

Exclusion Criteria:

* Pregnancy or lactation;
* Patients have aminoglycosides or vit B12.
* Prior BTX-A treatment to the masseter within the previous 12 months;
* Neuromuscular disorders or hypersensitivity to BTX-A or zinc compounds;
* Systemic illness affecting zinc metabolism (e.g., hepatic, renal, or metabolic disorders);
* Active infection, inflammation, or cutaneous lesions at the injection site.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome | 12 weeks
  • Percentage change in surface electromyographic (sEMG) amplitude of the masseter muscle at 12 weeks post-injection compared with baseline (normalized to maximal voluntary clench [MVC]).
  This endpoint captures the magnitude and persistence of neuromuscular inhibition, corresponding to the clinically relevant window where BTX-A efficacy typically begins to wane.

SECONDARY OUTCOMES:
Secondary Outcome | 12 weeks
  • Patient satisfaction (5-point likert scale);

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Asmi, Study Chair — lattakia university
Locations (1):
- lattakia University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Effect of zinc or copper supplementation on the efficacy and sustainability of botulinum toxin A "Botox" injection in masseter muscle of albino rats — https://doi.org/10.1016/j.jormas.2024.102156
- See also: Effects of zinc supplementation on duration and action of botulinum toxin applied to face muscles: A systematic review of randomized clinical trials — https://doi.org/10.1016/j.jtemin.2023.100080
- See also: Botulinum toxin type A injections for masticatory muscles hypertrophy: A systematic review — https://pubmed.ncbi.nlm.nih.gov/34620536/